CLINICAL TRIAL: NCT07287410
Title: Dementia and Mild Cognitive Impairment: Assessment of Cognitive Functioning, Functional Autonomy, and Neuropsychiatric Symptoms.
Acronym: RE-MIDA
Status: Recruiting | Type: Observational
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Principal Investigator, Francesco Corallo, Psychological manager, IRCCS Centro Neurolesi Bonino Pulejo
Other Study IDs: 20/2025
Record Dates: First submitted 2025-11-21; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Dementia; Mild Cognitive Impairment (MCI)
Keywords: Dementia; Mild Cognitive Impairment; neuropsychological; Activities of Daily Living; Neuropsychiatric symptoms
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: none - observational study — none - observational study

SUMMARY:
Dementia, in its various forms, is characterized by a generalized cognitive decline that can significantly compromise personal autonomy and quality of life. Mild Cognitive Impairment (MCI), although not classified as an overt form of dementia, represents a condition at evolutionary risk and is considered a crucial transitional stage for the early detection of cognitive decline. Understanding the impact of dementia and MCI from a multidimensional perspective is now essential to fully grasp the repercussions of these conditions on patients' daily lives. The present protocol aims to investigate key aspects related to these disorders, with the objective of exploring cognitive functioning, the degree of impairment in activities of daily living, and the presence of neuropsychiatric symptoms. Through an integrated and multidisciplinary approach, the study seeks to enhance clinical management and patient care, promoting more effective, targeted, and personalized interventions.

DETAILED DESCRIPTION:
The present protocol aims to evaluate several fundamental aspects related to dementia and Mild Cognitive Impairment (MCI). Specifically, the objective is to investigate cognitive functioning, the degree of impairment in autonomy in activities of daily living, and the presence of neuropsychiatric and mood disorders. Through this integrated perspective, the study seeks to promote improvements in clinical management and patient care, fostering more effective and personalized interventions. The primary objective of the study is to assess the level of functional autonomy in individuals affected by dementia or Mild Cognitive Impairment (MCI), with particular attention to both basic and instrumental activities of daily living, using the ADL and IADL scales. In addition to the main goal, the study aims to analyze the presence and extent of emotional and neuropsychiatric symptoms and to evaluate their impact on the overall psychological well-being of patients, using standardized psychometric tools that will be described in detail in later sections.

The study has an observational, retrospective design. Data will be collected from the neuropsychological assessments of patients who have undergone at least three testing sessions, approximately 12 months apart, at the Neuropsychology Outpatient Clinic of the IRCCS Centro Neurolesi Bonino Pulejo.

The sample size estimation was conducted in relation to the primary objective-evaluating the level of functional autonomy impairment in patients diagnosed with dementia or MCI, measured using the ADL and IADL scales. It was hypothesized that a mean difference of at least 1 point on the IADL scale between the two groups (patients with dementia vs. patients with MCI) would be clinically significant, assuming a standard deviation of 1.5, based on literature and clinical practice data. The statistical power was calculated using the G*Power software (version 3.1), selecting a two-tailed independent-samples t-test. Assuming an effect size (d) of 0.5, a significance level (α) of 0.05, and a statistical power (1-β) of 80%, the calculation indicated that at least 64 participants per group (MCI and dementia) would be required, for a total of 128 participants. Considering a potential dropout or loss to follow-up rate of 15%, an overall recruitment target of approximately 151 patients has been set. Participants will be recruited from the Neuropsychology Outpatient Clinic of the IRCCS Centro Neurolesi Bonino Pulejo in Messina.

Participants will be included in the study if, based on the available clinical documentation, they meet the following criteria:

* Age between 50 and 86 years;
* Suspected or confirmed diagnosis of dementia or Mild Cognitive Impairment (MCI), referred to the Neuropsychology Clinic for an initial evaluation or clinical monitoring;
* Absence of behavioral, psychiatric, or sensory disturbances severe enough to significantly compromise the performance of cognitive tests or the completion of questionnaires.

Participants will be excluded from the study if, based on clinical record review, they meet any of the following conditions:

* Presence of neurological disorders other than dementia or MCI, such as recent stroke, severe traumatic brain injury, epilepsy, multiple sclerosis, or other atypical neurodegenerative diseases;
* Unstable major psychiatric comorbidities at the time of assessment (e.g., schizophrenia, bipolar disorder in the active phase, untreated severe depression);
* Severe uncorrected sensory deficits (visual or auditory) that compromise the validity of cognitive and functional assessments;
* Use of medications with a significant cognitive impact (e.g., sedatives, high-dose antipsychotics) not stabilized at the time of assessment;
* Presence of terminal medical or oncological conditions, or other diseases that have significantly interfered with the assessment procedures.

The study involves retrospective collection of clinical and functional data from patients diagnosed with dementia or Mild Cognitive Impairment (MCI). Data from standardized tests will be extracted and analyzed from the medical records and databases available at the Neuropsychology Outpatient Clinic of the IRCCS Centro Neurolesi Bonino Pulejo in Messina, without any direct interventions involving the patients. Data will be entered into a secure database accessible only to study collaborators via personal credentials.

The following data will be collected:

* Information necessary for retrospective verification of inclusion and exclusion criteria;
* Demographic and clinical history data, including information on disease history and comorbidities;
* Results from psychological, neuropsychological, and clinical tests administered during visits, including:

  * Mini-Mental State Examination (MMSE)
  * Montreal Cognitive Assessment (MoCA)
  * Milan Overall Dementia Assessment (MODA)
  * Activities of Daily Living / Instrumental Activities of Daily Living (ADL/IADL)
  * Beck Depression Inventory (BDI)
  * Beck Anxiety Inventory (BAI)
  * Geriatric Depression Scale (GDS)
  * Frontal Assessment Battery (FAB)
  * Hamilton Depression Rating Scale (HDR-S)
  * Hamilton Rating Scale for Anxiety (HRSA)
  * Clock Drawing Test (CDT)
  * Neuropsychiatric Inventory (NPI) This retrospective design allows for an in-depth analysis of disease progression and serves as a useful tool for the early identification of potential predictive factors of deterioration. The results are expected to have relevant implications for clinical management, intervention planning, and the personalization of patient care pathways.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 86 years.
* Suspected or confirmed diagnosis of dementia or mild cognitive impairment (MCI).
* Referral to the neuropsychology clinic for initial assessment or clinical monitoring.
* Absence of behavioral, psychiatric, or sensory disorders severe enough to significantly impair cognitive testing or completion of questionnaires.

Exclusion Criteria:

* Presence of neurological disorders other than dementia or MCI (e.g., recent stroke, severe traumatic brain injury, epilepsy, multiple sclerosis, atypical neurodegenerative diseases).
* Unstable major psychiatric comorbidities at the time of assessment (e.g., schizophrenia, bipolar disorder in active phase, untreated severe depression).
* Uncorrected severe sensory deficits (visual or auditory) affecting the validity of cognitive or functional assessments.
* Use of medications with significant cognitive impact (e.g., sedatives, high-dose antipsychotics) not stabilized at the time of evaluation.
* Presence of terminal medical or oncological conditions or other illnesses significantly interfering with the assessment procedures.

Ages: 50 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 151
Sampling Method: Probability Sample
Enrollment: 151 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Dementia or Mild Cognitive Impairment (MCI) with ADL | 12 MONTHS
  The primary outcome variable considered for calculation is the score of the Activities of Daily Living (ADL) scale, used as the main index of functional autonomy in subjects with dementia or mild cognitive impairment (MCI).

SECONDARY OUTCOMES:
Functional autonomy in instrumental activities measured with the Instrumental Activities of Daily Living (IADL) scale | 12 MONTHS
  Assessment of functional autonomy in instrumental activities of daily living in subjects with dementia or mild cognitive impairment (MCI) using the Instrumental Activities of Daily Living (IADL) scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Centro Neurolesi Bonino Pulejo, Messina, ME, Italy

IPD SHARING:
Plan to Share IPD: No